CLINICAL TRIAL: NCT05788380
Title: The Effect of Regular Exercising on Shoulder Pain and Scapular Endurance
Brief Title: Shoulder Pain and Scapular Endurance
Acronym: SME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, research assistant, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MUŞALPARSLAN
Record Dates: First submitted 2023-03-14; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Musculoskeletal Pain Disorder; Sport Injury
Keywords: Scapular Muscle Endurance; Shoulder Pain; Regular Exercising; Exercising
MeSH Terms: conditions — Collagen Diseases; Shoulder Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: In total, 200 individuals aged between 17-25 years, who had no neurological and orthopedic problems participated. Individuals who had surgical stabilization, previous shoulder complex fractures, positive impingement test results, and systemic diseases were excluded. Participants were categorized into the Regular Exercising (n = 100) and Sedentary (n = 100) Groups. The young adults who were using the fitness center by their preference (unprofessional), and who were regularly exercising, were included in the Regular Exercising Group. The volunteer young adults who were not exercising were included in the Sedentary Group. All participants gave written-informed consent before participation, and the study protocol conformed to the standards for human experiments set by the Declaration of Helsinki and was approved by Ethics Committee for Human Investigations of Mustafa Kemal University Ethics Committee (4298783/05022/4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Scapular Muscles Endurance (SME (Other): The Scapular Muscles Endurance (SME) test was used to assess the endurance of the Serratus Anterior muscles.
  Interventions: Other: EXERCİSE
- Vizual Analog Scale (Other): The VAS for pain, measures pain severity in the affected shoulder from 0 to 10 points, with 0 points representing no pain at all and 10 points representing pain as bad as it can be
  Interventions: Other: EXERCİSE

INTERVENTIONS:
Other: EXERCİSE — EXERCISE FOR HEALTH AND PAIN IMPROVEMENT

SUMMARY:
Objective: This study aimed to investigate the effects of regular exercising on scapular muscle endurance and shoulder pain in young individuals.

Methods: Participants' clinical and sociodemographic properties recorded, scapular muscle endurance assessed with Scapular Muscular Endurance (SME) test, and shoulder pain severity questioned using the Visual Analogue Scale.

DETAILED DESCRIPTION:
Background: Serratus Anterior and Trapezius muscles are the most important stabilizers of the scapulothoracic joint. The inadequate endurance of these muscles plays an important role in the decreased neuromuscular performance.

Objective: This study aimed to investigate the effects of regular exercising on scapular muscle endurance and shoulder pain in young individuals.

Methods: Participants' clinical and sociodemographic properties recorded, scapular muscle endurance assessed with Scapular Muscular Endurance (SME) test, and shoulder pain severity questioned using the Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

for exercise group;

* between 17-25 years ages
* who were using the fitness center by their preference (not professional)
* had active sporting life (not professional)
* who were regularly exercising

for sedentary group;

* between 17-25 years ages
* who had sedentary life style

Exclusion Criteria:

for boths group;

* Individuals who had surgical stabilization,
* who had previous shoulder complex fractures
* who had positive impingement test results
* who had systemic diseases
* who had neurological and orthopedic problems

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
The Scapular Muscles Endurance (SME) test | Evaluation was done at the first meeting with the participants.
  The Scapular Muscles Endurance (SME) test was used to assess the endurance of the Serratus Anterior muscles. For this test, the participant stood against the wall with their shoulders and elbows flexed to 900. There was no contact between the participant's arms and the wall. The subjects then held a green elastic exercise band (with a resistance of 2.3 kg, when stretched 100%), and an adjustable ruler was placed between their elbows to maintain the test position. While both scapulae were neutrally positioned, the participant was then asked to externally rotate the shoulders and to maintain this force for as long as they could hold and the holding duration was recorded in second. The test was ended when the participant was unable to maintain the resistance and dropped the adjustable ruler, failed to maintain 900 of shoulder flexion, or reported an unacceptable increase in discomfort (Edmondston et al. 2008).
Vizual Analog Scale | Evaluation was done at the first meeting with the participants.
  measures pain severity in the affected shoulder from 0 to 10 points, with 0 points representing no pain at all and 10 points representing pain as bad as it can be

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer çetişli korkmaz, Prof. Dr., Study Director — Pamukkale University; Esra Doğru HUZMELİ, Assoc Prof, Study Chair — Mustafa kemalU
Locations (1):
- Aziz Dengiz, Denizli, Pamukkale, Turkey (Türkiye)